CLINICAL TRIAL: NCT02393287
Title: Activity and Toxicity Profile of Eribulin Mesylate in Pretreated Metastatic Breast Cancer: an Observational Multicentric Retroprospective Study
Brief Title: Retroprospective Real Life Observatory of Eribulin
Acronym: ReProLine
Status: Completed | Type: Observational
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Other Study IDs: ICO-A-RSD-2014-07
Record Dates: First submitted 2015-02-04; First posted 2015-03-19 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Reproline: this is an observational trial ; there is no intervention
  Interventions: Other: Eribulin (ReProLine)

INTERVENTIONS:
Other: Eribulin (ReProLine) — this is an observational trial ; there is no intervention

SUMMARY:
The objective of this observatory is to evaluate the effecacy of Eribulin in patients with metastatic breast cancer on a recent prescription period.

Part of the data collection will be retrospective and the other part will be prospective for patients started treatment by Eribulin between November 2014 and September 2015. It will allow a better assessment on the safety profile of this drug.

DETAILED DESCRIPTION:
Approximately one third of patients treated for localized breast cancer will present a metastatic evolution and 5% of patients are metastatic immediately.

At this stage, the malignancy is incurable with a median survival from 2 to 3 years.

Metastatic breast cancer treatment is part of a multidisciplinary approach. These two objectives are to prolong survival and improve quality of life. At present, there is no standard after the first line of chemotherapy, with fe strategy studies Eribulin is now a new therapeutic option to consider. Many patients have benefited from this treatment option and it seems interesting to evaluate in real life the effecacy and tolerance of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patient with breast cancer, histologically proven, metastatic or locally advanced
3. Patient treated by Eribulin between January and October 2014 (for the retrospective part) or between November 2014 and September 2015 (for the prospective part).
4. Patient with at least an assessment of the response to Eribulin

Exclusion Criteria:

1. Presence of other neoplasia
2. Man

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population includes all patients treated by Eribulin for breast cancer whose treatment has been starting between January 2014 and September 2015
Sampling Method: Probability Sample
Enrollment: 753 (Actual)
Dates: Start 2014-11; Primary Completion 2016-09 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 1 year
  Overall survival is defined as the time between the first administration of Eribulin and death from any cause.

SECONDARY OUTCOMES:
Overall Survival by subgroup | 1 year
  Overall survival is defined as the time between the first administration of Eribulin and death from any cause in the following subgroups:
  * According to the administration line of Eribulin: administration in third line or more versus administration in first or second line or for locally advanced cancer,
  * in HER2 + population
  * in triple negative population
  * in the elderly (> 70 years)
  * in the overweight population (BMI> 30)
Progression free survival | 1 year
  Progression-free survival is defined as the time between the first administration of Eribulin and the first demonstrated progression by image
Treatment response rate | 1 year
  Treatment response rate will be assessed by:
  * the best response obtained between the first administration of treatment with Eribulin and demonstrated progression by image (according to RECIST 1.1 criteria) or clinical
  * the clinical benefit (number of complete responses, partial responses or persistent stabilities mare than 6 months).
Treatment's tolerance | 1 year
  The treatment's tolerance will be assessed by collecting adverse events ≥ grade 3 quoted according to NCI CTCAE v4.0 classification.

CONTACTS AND LOCATIONS:
Overall Officials: Anne PATSOURIS, MD, Principal Investigator — Institut de Cancerologie de l'Ouest
Locations (13):
- France (13):
  - Institut de Cancerologie de l'Ouest, Angers
  - CHU Jean Minjoz, Besançon
  - CHU, Brest
  - Centre Jean Bernard, Le Mans
  - Centre Léon Berard, Lyon
  - Institut de Cancerologie de l'Ouest, Nantes
  - Centre Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - CH, St-Malo
  - Centre Paul Strauss, Strasbourg
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy